CLINICAL TRIAL: NCT05575349
Title: Effects of Mandala Coloring on Anxiety and Quality of Life of Women in the Climacteric Period: Randomized Controlled Experimental Study
Brief Title: Effects of Mandala Coloring on Anxiety and Quality of Life of Women in the Climacteric Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Collaborators: Cukurova University (Other)
Responsible Party: Principal Investigator, Ayca Solt Kirca, Assistant Professor, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KırklareliED-1
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Anxiety; Climactericum
Keywords: Climacterium; Anxiety; Quality of life; Mandala coloring
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandala coloring group (Experimental): Mandala painting will be applied to climacteric women with anxiety.
  Interventions: Other: Mandala coloring
- Control group (No Intervention): Participants in this group will consist of people who do not routinely do any practice on their own to reduce anxiety symptoms

INTERVENTIONS:
Other: Mandala coloring — Participants will be asked to choose the pages they want from 12 colored felt-tip pen paint sets and 12 mandala coloring pages given to each participant by the researcher for 6 weeks, 1 days a week, at any time of the day and for an average of 20-30 minutes each time, and paint them in the colors they want.
  Arms: Mandala coloring group

SUMMARY:
This research was planned as a randomized controlled experimental study in order to reduce the anxiety felt and improve the quality of life by women in the climacteric period.

DETAILED DESCRIPTION:
Climacteric period; It is a life process in which the ovarian hormone and activity ends with a decrease, and the transition from the reproductive period to the non-reproductive period takes place, and includes perimenopause, menopause and postmenopausal stages. During the menopausal transition period, women experience many physical and psychological symptoms such as vasomotor symptoms, sleep disorders, depressed mood, and stress that negatively affect their quality of life. When the literature is examined, it can be seen that these menopausal symptoms experienced by women affect and trigger anxiety. Effective management of anxiety, which can negatively affect psychosocial well-being, social relations and mood, trigger or exacerbate menopausal symptoms, can improve the quality of life of women in the climacteric period. Therefore, anxiety management can be effective for women to cope with menopausal symptoms.

Carl Gustav Jung, a Swiss psychiatrist, discovered the therapeutic effect of coloring mandala, which is one of the art therapy methods in reducing anxiety. When the studies are examined, there have been many studies investigating the effect of Mandala coloring on reducing anxiety. Curry and Kasser (2005), Van der Vennet and Serice (2012), Flet et al (2017) stated that coloring mandala reduces anxiety on students; Gürcan and Atay Turhan (2021) and Yakar et al (2021) found that it reduces anxiety and depression in cancer patients; Khademi et al (2021) reported that it reduced anxiety in hospitalized covid-19 patients; Amelia et al (2020) found that it reduced anxiety in pregnant women.

When the studies are examined, there are studies showing that coloring mandala reduces anxiety in cancer patients, children, and pregnant women, but no study has been found on the effect of reducing anxiety related to menopausal symptoms and improving the quality of life of women in the climacteric period. This research was planned as a randomized controlled experimental study in order to reduce the anxiety felt and improve the quality of life by women in the climacteric period.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Fully answering survey and scale forms.
* Ability to read and understand Turkish
* Being in the climacteric period (42-65 years)
* Having 40 or more from STAI

Exclusion Criteria:

* Unwilling to continue working
* Having any problem that prevents communication (such as hearing, speaking, and understanding abilities),
* Taking medication for menopausal symptoms
* Using one of the pharmacological or non-pharmacological methods to reduce anxiety and receiving psychiatric treatment (Pharmacotherapy or psychotherapy).
* Surgical menopause
* Having a mental illness

Ages: 42 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 80 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-06-17 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form | between one to six months
  A form that includes questions about women's socio-demographic and menopausal and characteristics.

SECONDARY OUTCOMES:
the Spielberger State-Trait Anxiety Inventory (STAI) Scale | between one to six months
  This scale, developed by Spielberg in 1973, consists of 20 questions. It is a 4-point Likert type scale (1=not at all, 4=very much). The lowest score that can be obtained from the scale is 20, and the highest score is 80. The higher the score is, the higher the anxiety level is. The alpha value of the scale is 0.86-.92.33. The validity and reliability study in our country was conducted by Oner et al., in 1983 and the alpha value was found between 0,83 and 0,87. The scale that will be used to evaluate the state and trait anxiety of pregnant women. As the score increases, it is determined that the anxiety is higher.

OTHER OUTCOMES:
Menopause-Specific Quality of Life Questionnaire | between one to six months
  This scale was developed by Hilditch, Lewis et al. in 1996 to create a health-specific quality of life scale in menopause with psychometric properties based on women's experiences. It was adapted to Turkish society by Kharbouch and Sahin in 2005 and its validity and reliability were determined. It consists of 29 questions and each sub-domain score is ordered from 1 to 8. As the score increases, the severity of the complaint also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Ayça ŞOLT KIRCA, Principal Investigator — Kırklareli University; Efsun DERIN, Study Director — Kırklareli University; ELIF DAGLI, Study Director — Cukurova University
Locations (1):
- Kırklareli Training and Research Hospital, Kırklareli, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No